CLINICAL TRIAL: NCT03620864
Title: Motor Control Exercises and Neurodynamic Intervention for Lumbar Radiculopathy: A Randomized Clinical Trial
Brief Title: Neurodynamic Intervention for Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Director, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HU201531
Record Dates: First submitted 2018-07-24; First posted 2018-08-08 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor control exercise (Active Comparator): Patients will receive 8 sessions of motor control exercise program of 30 min duration for 4 weeks, twice per week. Exercises will be demonstrated to the participants by an experienced physical therapist. On each session, the therapist will correct each subject personally. Participants will be asked for practicing the exercises at home once daily for 20 minutes over the 8-week intervention period. The motor control exercise program will consist of a progression from isolated contraction of the transversus abdominis and/or isolated contraction of the multifidi to combined contraction of both transversus abdominis in different positions from supine or prone to bridging or four-point kneeling.
  Interventions: Other: Motor Control Exercises
- Motor control exercise plus neurodynamic intervention (Experimental): Patients will receive 8 sessions of motor control exercise program of 30 min duration for 4 weeks, twice per week. Exercises will be demonstrated to the participants by an experienced physical therapist. On each session, the therapist will correct each subject personally. Participants will be asked for practicing the exercises at home once daily for 20 minutes over the 8-week intervention period. The motor control exercise program will consist of a progression from isolated contraction of the transversus abdominis and/or isolated contraction of the multifidi to combined contraction of both transversus abdominis in different positions from supine or prone to bridging or four-point kneeling. In addition, participants allocated to the neurodynamic group will also receive a nerve neurodynamic slider intervention targeting the main trunk of the sciatic nerve of the affected side during al treatment sessions (n=8).
  Interventions: Other: Motor Control Exercise Plus Neurodynamic Intervention

INTERVENTIONS:
Other: Motor Control Exercises — Patients will receive 8 sessions of motor control exercise program of 30 min duration for 4 weeks, twice per week. Exercises will be demonstrated to the participants by an experienced physical therapist. On each session, the therapist will correct each subject personally. Participants will be asked for practicing the exercises at home once daily for 20 minutes over the 8-week intervention period. The motor control exercise program will consist of a progression from isolated contraction of the transversus abdominis and/or isolated contraction of the multifidi to combined contraction of both transversus abdominis in different positions from supine or prone to bridging or four-point kneeling.
  Arms: Motor control exercise
Other: Motor Control Exercise Plus Neurodynamic Intervention — Patients will receive 8 sessions of motor control exercise program of 30 min duration for 4 weeks, twice per week. Exercises will be demonstrated to the participants by an experienced physical therapist. On each session, the therapist will correct each subject personally. Participants will be asked for practicing the exercises at home once daily for 20 minutes over the 8-week intervention period. The motor control exercise program will consist of a progression from isolated contraction of the transversus abdominis and/or isolated contraction of the multifidi to combined contraction of both transversus abdominis in different positions from supine or prone to bridging or four-point kneeling. In addition, participants allocated to the neurodynamic group will also receive a nerve neurodynamic slider intervention targeting the main trunk of the sciatic nerve of the affected side during al treatment sessions (n=8).
  Arms: Motor control exercise plus neurodynamic intervention

SUMMARY:
Low back pain (LBP) is a common condition and has a significant impact on the individual in terms of pain and disability. Lumbar radiculopathy occurs often with LBP and may be the result of a lumbar herniated disc which will irritate a lumbar nerve trunk resulting in intraneural inflammation. There is evidence supporting the use of manual therapies of lumbar radiculopathy. One potential manual therapy is neurodynamic mobilization technique. No scientific evidence, based on a RCT, exists that this particular approach is beneficial for individuals with LBP and lumbar radiculopathy

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a confirmed (via MRI) disc herniation at between L4 and S1 level;
* Subjects exhibiting lumbar radiating pain in the lower extremity for at least 3 months
* Subjects with a positive straight leg raise with symptoms reproduction

Exclusion Criteria:

* indication for surgical intervention;
* had a confirmed disc herniation at other lumbar levels;
* have had any other spinal conditions such as spinal tumors or spondylolisthesis;
* had received treatment for this condition by a physical therapist the previous 6 month;
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Changes in Lower Extremity Pain Intensity | Baseline, after 4 treatment sessions, after 8 treatment sessions,and 2 months after last treatment session
  A Numerical Pain Rate Scale (NPRS, 0-10) where 0 represents no pain and 10 the maximum pain will be used to record the mean intensity of pain in the lower extremity

SECONDARY OUTCOMES:
Changes in Neuropathic Mechanism Consideration | Baseline, after 4 treatment sessions, after 8 treatment sessions,and 2 months after last treatment session
  The Self-report Leeds Assessment of Neuropathic Symptoms and Signs Scale (S-LANSS) will be used for assessing neuropathic mechanism. The S-LANSS is a 7-item tool for identifying patients whose pain is dominated by neuropathic mechanisms. Each item is a binary response (yes or no) to the presence of symptoms (5 items) or clinical signs (2 items). The total score is 24 points and a value ≥ 12 points is indicative of a neuropathic component of pain.
Changes in Related-Disability | Baseline, after 4 treatment sessions, after 8 treatment sessions,and 2 months after last treatment session
  The Roland-Morris Disability Questionnaire will be used for assessing related-disability. The score can range from 0-24 with higher scores indicative of higher related-disability.
Changes in Mechanical Sensitivity of the Sciatic Nerve | Baseline, after 4 treatment sessions, after 8 treatment sessions,and 2 months after last treatment session
  The degrees of the straight leg raise test will be used to assess sensitivity of the sciatic nerve
Changes in Pressure Pain Thresholds | Baseline, after 4 treatment sessions, after 8 treatment sessions,and 2 months after last treatment session
  Pressure pain thresholds will be assessed with a mechanical algometer over the common peroneal and tibial nerve

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

REFERENCES:
- [Derived] Plaza-Manzano G, Cancela-Cilleruelo I, Fernandez-de-Las-Penas C, Cleland JA, Arias-Buria JL, Thoomes-de-Graaf M, Ortega-Santiago R. Effects of Adding a Neurodynamic Mobilization to Motor Control Training in Patients With Lumbar Radiculopathy Due to Disc Herniation: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2020 Feb;99(2):124-132. doi: 10.1097/PHM.0000000000001295. PMID 31464753